CLINICAL TRIAL: NCT03585127
Title: A Pilot Randomized Controlled Study to Compare Avatar Therapy and Cognitive Behavioral Therapy in Patients With Treatment-resistant Schizophrenia.
Brief Title: Avatar Therapy in Comparison to Cognitive Behavioral Therapy for Treatment-resistant Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Otsuka Canada Pharmaceutical Inc. (Industry)
Responsible Party: Principal Investigator, Alexandre Dumais, Psychiatrist, Clinical Associate Professor, Principal Investigator, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPPM 16-17 - 06
Record Dates: First submitted 2018-07-02; First posted 2018-07-12 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Auditory Hallucination, Verbal; Treatment-resistant Schizophrenia
Keywords: Auditory verbal hallucinations; Schizophrenia; Treatment-resistant; Psychotherapy; Cognitive Behavioral Therapy; Avatar Therapy; Virtual reality
MeSH Terms: conditions — Hallucinations; Schizophrenia, Treatment-Resistant; Schizophrenia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy comprises of nine weekly sessions of an hour.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Avatar Therapy (Experimental): Avatar Therapy consists of 9 weekly sessions: one avatar creation session and 8 therapeutic sessions of one hour.
  Interventions: Behavioral: Avatar Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will be offered 9 individual and weekly sessions of 1 hour, which will be administered in an individual format by a licensed psychologist or psychiatrist trained in Cognitive Behavioral Therapy for psychosis (CBTp). The program is derived and adapted from current evidence-based treatments for hallucinations. The 9 CBTp sessions will consist of a succession of learning modules and suggested task assignments.
  Other Names: CBT for psychosis
  Arms: Cognitive Behavioral Therapy
Behavioral: Avatar Therapy — Participants will be offered 9 individual and weekly sessions of 1 hour, which will be administered in an individual format by a licensed psychologist or psychiatrist experienced with psychosis patients. The therapy will consist in prompting participants to enter in a dialogue with their persecutor to better regulate their emotional responses. Over the course of the therapy, the avatar's speech and tone will gradually be changed by the therapist to echo participants' improved ability to regulate their emotions. That is, the avatar will progressively change from being abusive to becoming helpful and supportive. By doing so, the therapy will seek to reinforce participants' feeling of empowerment over their voices.
  Arms: Avatar Therapy

SUMMARY:
Schizophrenia is associated with long-lasting health, social and financial burden for patients, families, caregivers and society. Unfortunately, 25-30% of schizophrenia patients respond poorly to antipsychotic medication. Moreover, psychotherapeutic treatment alternatives are very limited for this suffering population. This unmet clinical need requires innovation and action. Psychotherapeutic treatment alternatives such as Cognitive Behavior Therapy (CBT) provide at best moderate results. Using immersive virtual reality, we recently tested a novel psychotherapeutic intervention, Avatar Therapy (AT), where the therapist engages in a dialogue with the patient through a virtual representation of the patient's distressing voice. This approach, being both relational and experiential, provides a unique opportunity to aid patients gain control over their voice. The results of our pilot study on AT were clinically promising for the severity and distress related to hallucinations, positive symptomatology and emotion regulation. To further research in this field, the primary goal of this randomized-controlled, single-site parallel study is to show that AT is superior to CBT for the treatment of persistent auditory hallucinations in schizophrenia. Our secondary goal is to examine the effects of these interventions on emotion regulation, mood symptoms (anxiety and depression), self-esteem, level of functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* distressing auditory verbal hallucinations
* medication resistance relating to auditory verbal hallucinations (no response after 3 antipsychotics trials lasting at least 4 weeks each with a minimum of 400mg chlorpromazine equivalent)
* DSM-5 diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* any change in medication within the past 2 months;
* substance use disorder within the last 12 months
* neurological disorder or unstable and serious physical illness
* ongoing psychotic episode
* Cognitive Behavioral Therapy for psychosis within the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Psychotic Symptom Rating Scale (PSYRATS) - auditory hallucinations | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  11-item structured interview assessing the severity of auditory hallucinations; Range 0-44, Higher values indicate a worse outcome

SECONDARY OUTCOMES:
Change in Beliefs About Voices Questionnaire - Revised (BAVQ-R) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  35-item self-reported measure designed to assess key beliefs and responses people have concerning their voice; Range 0-105, Higher scores indicate more beliefs and responses toward their voice
Change in Positive And Negative Syndrome Scale (PANSS) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  30-item semi-structured interview investigating overall symptoms severity of schizophrenia in the last week; Range 30-210, Higher values indicate a more severe symptomatology
Change in Beck Depression Inventory - II (BDI-II) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  21-item self-reported measure assessing depression symptoms over the past 2 weeks; Range 0-63, Higher values indicate more severe depressive symptomatology
Change in Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (QLESQ-SF) | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  16-item self-reported scale measuring enjoyment and satisfaction experienced during the past week in various areas of daily functioning; Range 14-70, Higher values indicate a better satisfaction of life
Change in Empowerment scale (Making Decisions) - Revised Short Form | Within 1 week before treatment, within 1 week after treatment, follow-ups at 3 months, 6 months and 12 months
  25-item self-reported scale measuring the feeling of empowerment; Range 25-100, Higher values indicate a stronger feeling of empowerment

OTHER OUTCOMES:
Change in Igroup Presence Questionnaire (IPQ) | At the end of each Avatar Therapy session
  14-item scale measuring the sense of presence; Range 0-84, Higher values indicate a stronger feeling of presence

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Dumais, MD, Ph.D, Principal Investigator — Institut Philippe Pinel de Montréal
Locations (1):
- Institut Universitaire en Santé Mentale de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hudon A, Leveille N, Sanchez-Schicharew K, Dellazizzo L, Phraxayavong K, Dumais A. The impacts of the COVID-19 pandemic on treatment-resistant schizophrenia patients having followed virtual reality therapy or cognitive behavioural therapy: a content analysis. Ann Med. 2022 Dec;54(1):2477-2485. doi: 10.1080/07853890.2022.2121852. PMID 36102593